CLINICAL TRIAL: NCT03865888
Title: Evaluation of the Effect of Topical Application of Tacrolimus 0.03% (FK506) Eye Drops Versus Cyclosporine 0.05% Eye Drops in Treatment of Dry Eye in Secondary Sjogren Syndrome
Brief Title: Comparing Effect of Topical Tacrolimus 0.03% Versus Cyclosporine 0.05% in Dry Eyes of Secondary Sjogren Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pavly Moawd (Other)
Responsible Party: Sponsor-Investigator, Pavly Moawd, Assistant Lecturer of Ophthalmic Medicine and Surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-75-2018
Record Dates: First submitted 2018-12-16; First posted 2019-03-07 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye; Sjogren Syndrome
Keywords: Sjogren Syndrome; Dry eye; Cyclosporine; Tacrolimus
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome | interventions — Cyclosporins; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Evaluation of the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops in treatment of dry eye in Secondary Sjogren Syndrome.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporins 0.05 % treated eyes (Active Comparator): Topical Cyclosporins 0.05% eye drops twice in one eye for 3 months
  Interventions: Drug: Cyclosporins
- Tacrolimus 0.03% treated eyes (Active Comparator): Topical Tacrolimus 0.03% eye drops twice in one eye for 3 months
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporins — Cyclosporins eye drops to be administered in dry eyes
  Other Names: Restasis
  Arms: Cyclosporins 0.05 % treated eyes
Drug: Tacrolimus — Tacrolimus eye drops to be administered in dry eyes
  Other Names: FK506
  Arms: Tacrolimus 0.03% treated eyes

SUMMARY:
Evaluation of the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops in treatment of dry eye in Secondary Sjogren Syndrome.

DETAILED DESCRIPTION:
Sjogren syndrome is a chronic autoimmune disorder characterized by immune cell infiltration of exocrine glands (exocrinopathy or epitheliitis) and systemic complications due to autoantibody production, immune complex deposition and lymphocytic infiltration of many organs .The loss of aqueous tear flow in Sjogren syndrome is a result of inflammatory cell infiltration of the lacrimal glands.The principal ocular manifestation of which is decreased tear production leading to chronic irritation and damage to the corneal and conjunctival epithelium. Dry eye associated with Sjogren syndrome (SS dry eye) is often more severe than non-Sjogren dry eye (non-SS dry eye). Rose bengal staining, fluorescein staining, impression cytology, and brush cytology show greater changes in SS dry eye owing to a lack of both basic tearing and reflex tearing resulting from lacrimal gland destruction, which is the hallmark of deteriorating clinical conditions.

The initial tear film ocular surface society dry eye workshop report noted the importance of ocular surface inflammation not only in the development of, but as a downstream effect and propagator of dry eye disease , and reviewed a range of therapies that function, at least in part, by anti-inflammatory mechanisms of action. Thus understanding the link between inflammation and dry eye validates the utilization of anti-inflammatory therapy in everyday practice.

Cyclosporine is understood to be an immunomodulatory drug with anti-inflammatory properties, as well as having other actions relevant to managing dry eye disease . Topical cyclosporine was approved by the FDA for the treatment of moderate-to-severe dry eye disease in 2003, based on an improvement in tear production.

Tacrolimus, a macrolide produced by Streptomyces tsukubaensis,was discovered in 1984 in Japan while searching for new immunosuppressive and cancer chemotherapeutic agents. The use of tacrolimus is of special interest in ophthalmology because it is indicated to be effective in the treatment of immune-mediated diseases Thus, the investigators performed this study to evaluate the effect of two different immunomodulatory eye drops on the ocular surface which are topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops in treatment of dry eye in Secondary Sjogren Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as Secondary Sjogren syndrome according to the 2002 American European consensus group (AECG) criteria, which require the presence of well defined major connective tissue disease (such as rheumatoid arthritis and systemic lupus erythematosus.
* All patients show chronic symptoms of burning, foreign body sensation, itching in both eyes, abnormal Schirmer test <5 mm wetting of the paper after 5 minutes, and abnormal tear breakup time (TBUT) < 10 seconds.
* Wash out period of 30 days before start of the immunomodulatory eye drops included in the investigator's study

Exclusion Criteria:

1. Any inflammation or active structural changes in the iris or anterior chamber.
2. Patients receiving or who had received systemic cyclosporine or tacrolimus.
3. Patients receiving any systemic drug that can cause dry eye as some antidepressants , antihistaminic drugs , hormonal therapy…etc
4. Glaucoma.
5. Previous ocular surgery.
6. Use of any topical medication other than artificial tears.
7. Contact lens wearers.
8. Presence of any corneal infection.
9. Any corneal diseases (ulcer, opacity, scar, bullous keratopathy, symblepharon or tumors).
10. Deforming structural lid or conjunctival abnormality.
11. Pregnancy.
12. Prior diagnosis of any of the following conditions would exclude participation in AECG study :

Past head and neck radiation treatment Hepatitis C infection Acquired immunodeficiency disease (AIDS) Pre-existing lymphoma Sarcoidosis Graft versus host disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison between the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops on tear film volume in dry eyes in Secondary Sjogren Syndrome patients. | 3 months follow up
  Tear film volume will be evaluated using Schirmer I test in millimetres in seconds in dry eyes before and after prescribing either cyclosporine or tacrolimus eye drops in Secondary Sjogren Syndrome patients.
Evaluating the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops on ocular surface damage in dry eyes in Secondary Sjogren Syndrome patients. | 3 months follow up
  Ocular surface damage will be assessed in term of calculating ocular surface staining score in dry eyes of Secondary Sjogren Syndrome patients before start and at end of treatment in cyclosporine and tacrolimus treated eyes.
Studying the effect of cyclosporine and tacrolimus eye drops on tear film stability in dry eyes in Secondary Sjogren Syndrome patients. | 3 months follow up
  Tear film stability will be described in form of tear film break up time in seconds in treated dry eyes of Secondary Sjogren Syndrome patients before and after adminstration of cyclosporine and tacrolimus eye drops.

SECONDARY OUTCOMES:
Evaluating the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops on meibomian glands secretion in dry eyes of Secondary Sjogren Syndrome patients. | 3 months follow up
  Comparing between effect of topical cyclosporine 0.05% and tacrolimus 0.03 % on meibomian glands secretions quality score in dry eyes of Secondary Sjogren Syndrome patients.
Studying the effect of topical application of Tacrolimus 0.03% (FK506) eye drops versus Cyclosporine 0.05% eye drops on expressibility of meibomian glands in dry eyes of Secondary Sjogren Syndrome patients. | 3 months follow up
  Evaluating the effect of topical cyclosporine 0.05% and tacrolimus 0.03 % on meibomian glands expressibility score in dry eyes of Secondary Sjogren Syndrome patients.

CONTACTS AND LOCATIONS:
Overall Officials: Omar El Zawahry, Principal Investigator — Cairo University; Gaafar Ragab, Principal Investigator — Cairo University; Rehab Shamma, Principal Investigator — Cairo University
Locations (1):
- Pavly Moawad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moawad P, Shamma R, Hassanein D, Ragab G, El Zawahry O. Evaluation of the effect of topical tacrolimus 0.03% versus cyclosporine 0.05% in the treatment of dry eye secondary to Sjogren syndrome. Eur J Ophthalmol. 2022 Jan;32(1):673-679. doi: 10.1177/1120672121992680. Epub 2021 Feb 2. PMID 33530719